CLINICAL TRIAL: NCT02163109
Title: Measurement of Oxygen Consumption in Critical Illness Using Optical Gas Analysis
Brief Title: Oxygen Consumption in Critical Illness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 14/EE/0003
Record Dates: First submitted 2014-06-09; First posted 2014-06-13 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Critical Illness
Keywords: Oxygen consumption; Pulmonary gas exchange; Cardiac output
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically-ill patients: Adult patients requiring intubation and mechanical ventilation on an intensive care unit, predicted to require a further 48 hours of artificial ventilation

SUMMARY:
Many serious illnesses are characterised by a lack of oxygen delivery to the body's tissues. This can be due to problems with the circulation, such as when the heart fails to pump blood efficiently or if the blood pressure is very low, or due to changes in the lungs preventing them from transferring oxygen effectively from the air into the blood.

Many of the treatments used in critically ill patients are aimed at improving the supply of oxygen-rich blood to the tissues. These include drugs to increase the blood pressure or make the heart pump more forcibly, blood transfusions to increase the amount of oxygen that the blood can carry, and ventilators (breathing machines) to help the lungs introduce more oxygen into the bloodstream. Decisions to use such treatments are based on a number of factors. One of the most important is an assessment of how much oxygen an individual patient is using at a given time. Whilst it is possible to measure average oxygen consumption over a long period of time in healthy individuals, the equipment and techniques needed are simply not practical for routine use in the clinical setting of a critical care unit. Critical care doctors and nurses therefore have to rely on a number of different indicators of the adequacy of the amount of oxygen that is being provided in order to make decisions about how best to treat patients. Unfortunately, all of these have their limitations, are affected by other treatments patients may be receiving, and can be difficult to interpret. Examples include 'mixed venous oxygen saturation' (SvO2), that is the amount of oxygen in the blood coming back to the lungs from the body, ready to have more oxygen added, and blood lactate levels, which give an indication of whether the tissues have enough oxygen to produce the energy they need to function in an efficient manner.

Our group has developed a device which can be added easily to the normal equipment used on a critical care ward when a patient is on a ventilator, which can accurately and rapidly measure the amount of oxygen the individual is consuming.

This study will provide us with data so the investigators can define a "normal" range of oxygen consumption in these patients, and treatments which alter consumption. In a future study, once the investigators know what the normal range is, they can introduce new techniques to improve oxygen consumption in those patients whose consumption is less than ideal.

DETAILED DESCRIPTION:
This is a prospective longitudinal observational study in thirty intubated, ventilated patients. Patients will be recruited from the population of already intubated and ventilated individuals on an adult intensive care unit (AICU). Once patients have been recruited we will insert the optical gas analyser (OGA) into the ventilation circuit (tubing) for 48 hours.

Data will be continuously collected until 48 hours from attachment of the OGA, death or extubation of the patient, and analysed retrospectively. A time series describing oxygen consumption with a resolution of one minute or less will be prepared and standard measures of dispersion calculated. In addition, variables that are routinely recorded on the computerised clinical record during the same period will then be examined and associations sought between these variables and changes in oxygen consumption as measured with the OGA. We have prospectively identified variables which, based on the published literature, are likely to be associated with variation in oxygen consumption (VO2) upon which attention will focus, though others may become apparent during the study:

* Body temperature
* Seizures
* Change in haemoglobin concentration (including due to blood transfusion)
* Bolus fluids
* Vasoactive drugs
* Beta-agonist drugs
* Drugs affecting the angiotensin-converting enzyme system
* Renal replacement therapy
* Feeding
* Sedation
* Neuromuscular blockers
* Mode of ventilation
* Fraction of inspired oxygen (FiO2)
* Physical activity
* Surgery

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years or over
* Admitted to an adult intensive care unit
* Expected duration of intubation and mechanical ventilation of at least 48 hours

Exclusion Criteria:

* Consultee indicates patient would be likely to decline enrolment
* Patient is receiving palliative care
* Use of active cooling
* Heavy sputum production (or other indication) necessitating use of an active humidifier in ventilator circuit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients requiring intubation and mechanical ventilation on an adult intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption | Up to 48 hours
  Within patient oxygen consumption over time correlated with changes in physiological variables and treatment received

CONTACTS AND LOCATIONS:
Overall Officials: John D Young, DM, Principal Investigator — University of Oxford and Oxford University Hospitals NHS Trust
Locations (1):
- Oxford Univerity Hospital NHS Trust, John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Cummings B, Hamilton ML, Ciaffoni L, Pragnell TR, Peverall R, Ritchie GA, Hancock G, Robbins PA. Laser-based absorption spectroscopy as a technique for rapid in-line analysis of respired gas concentrations of O2 and CO2. J Appl Physiol (1985). 2011 Jul;111(1):303-7. doi: 10.1152/japplphysiol.00119.2011. Epub 2011 Apr 21. PMID 21512147
- [Background] Shoemaker WC, Appel PL, Kram HB. Hemodynamic and oxygen transport responses in survivors and nonsurvivors of high-risk surgery. Crit Care Med. 1993 Jul;21(7):977-90. doi: 10.1097/00003246-199307000-00010. PMID 8319478
- [Background] Hayes MA, Timmins AC, Yau EH, Palazzo M, Hinds CJ, Watson D. Elevation of systemic oxygen delivery in the treatment of critically ill patients. N Engl J Med. 1994 Jun 16;330(24):1717-22. doi: 10.1056/NEJM199406163302404. PMID 7993413
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] ProCESS Investigators; Yealy DM, Kellum JA, Huang DT, Barnato AE, Weissfeld LA, Pike F, Terndrup T, Wang HE, Hou PC, LoVecchio F, Filbin MR, Shapiro NI, Angus DC. A randomized trial of protocol-based care for early septic shock. N Engl J Med. 2014 May 1;370(18):1683-93. doi: 10.1056/NEJMoa1401602. Epub 2014 Mar 18. PMID 24635773
- [Background] Shoemaker WC, Appel PL, Kram HB, Waxman K, Lee TS. Prospective trial of supranormal values of survivors as therapeutic goals in high-risk surgical patients. Chest. 1988 Dec;94(6):1176-86. doi: 10.1378/chest.94.6.1176. PMID 3191758